CLINICAL TRIAL: NCT06672549
Title: A Master Protocol for a Randomized, Controlled, Clinical Platform Trial to Investigate the Efficacy and Safety of Interventions for Chronic Weight Management in Pediatric Participants With Obesity or Overweight
Brief Title: A Platform Trial for Pediatric Participants With Obesity or Overweight (LY900040)
Acronym: ADVANCE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18865; J4M-MC-PWMP (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — orforglipron

STUDY DESIGN:
Intervention Model Description: The PWMP protocol includes screening assessments plus a framework for the subsequent intervention, which is the primary purpose of the protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Orforglipron (ISA PW01) (Experimental): Participants will receive orforglipron or placebo orally. Each ISA will detail the intervention specific.
  Interventions: Drug: Orforglipron; Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally. ISA specific interventions will be listed in the ISA.
  Other Names: LY3502970
Drug: Placebo — Administered orally. ISA specific interventions will be listed in the ISA.

SUMMARY:
The purpose of this pediatric, chronic weight management, Phase 3 Master Protocol (PWMP) is to create a framework to evaluate the safety and efficacy of pharmacologic agents for the treatment of obesity or overweight in pediatric participants.

DETAILED DESCRIPTION:
The PWMP establishes entry criteria for newly enrolled participants across the master and the ISAs. The ISAs may start independently of other ISAs as interventions become available for clinical testing. PWMP results will be reported when all the ISA's complete.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of at least 1 unsuccessful effort to lose sufficient body weight after participation in a structured lifestyle modification program (diet and exercise counseling for at least 3 months) prior to screening.
* Obesity as defined by BMI equal to or above the 95th percentile for age and sex (on age- and gender-specific growth chart [CDC-NCHS, 2022]); OR
* Applies to participant age between 12 and <18 years old. Overweight as defined by BMI equal to or above the 85th percentile but less than the 95th percentile for age and sex, on age- and sex-specific growth chart (CDC-NCHS, 2022), and at least 1 weight-related comorbidity,

  * hypertension
  * type 2 diabetes (T2D)
  * prediabetes
  * dyslipidemia
  * obstructive sleep apnea
  * metabolic dysfunction-associated steatohepatitis (MASH) or metabolic dysfunction-associated steatotic liver disease (MASLD)

Exclusion Criteria:

* Have undergone or plan to undergo weight reduction procedure during the study, such as, but not limited to:

  * gastric bypass
  * sleeve gastrectomy
  * restrictive bariatric surgery, such as Lap-Band® gastric banding, or
  * any other procedure intended to result in weight reduction.
* Have a diagnosis that is a secondary cause of obesity or have a history of abrupt onset of obesity suggesting a secondary cause, such as hypothalamic, monogenetic, syndromic, or endocrine causes.
* Have a self-reported, or by parent or legal guardian where applicable, decrease in body weight greater than 5 kg (11 lbs) within 90 days before screening irrespective of medical records
* Have type 1 diabetes or history of ketoacidosis, or hyperosmolar state.
* Have HbA1c >9.0% (75 mmol/mol) as measured by central laboratory at screening.
* Have a family or personal history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia Syndrome Type 2.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Allocated to Each ISA | Baseline to Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (41):
- United States (16):
  - Carey Chronis MD Pediatric, Infant and Adolescent Medicine, Ventura, California
  - Yale School of Medicine - Yale Diabetes Center (YDC)) Trials, New Haven, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Children's Healthcare of Atlanta - Center for Advanced Pediatrics, Atlanta, Georgia
  - Ann and Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Velocity Clinical Research, Lafayette, Louisiana
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Gulfport, Mississippi
  - Sundance Clinical Research, St Louis, Missouri
  - Velocity Clinical Research, Omaha, Nebraska
  - Lucas Research, Inc, Morehead City, North Carolina
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Health One Hundred Oaks, Nashville, Tennessee
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Houston, Texas
  - La Providence Pediatrics Clinic - Chemidox Clinical Trials, Houston, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
- Brazil (3):
  - L2IP - Instituto de Pesquisas Clínicas, Brasília
  - Hospital Universitario de Caxias do Sul, Caxias do Sul
  - CPQuali Pesquisa Clínica Sao Paulo, São Paulo
- Israel (3):
  - Yitzhak Shamir Medical Center, Beer Yaacov
  - Shaare Zedek Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (4):
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- Mexico (4):
  - Centro Para el Desarrollo de la Medicina y de Asistencia Especializada SC, Culiacán
  - PanAmerican Clinical Research - Guadalajara, Guadalajara
  - Innovacion y Desarrollo de Estrategias en Salud SA de CV, Mexico City
  - Hospital Angeles Puebla, Puebla City
- Poland (4):
  - Krakowskie Centrum Medyczne, Krakow
  - Instytut Diabetologii, Warsaw
  - FutureMeds - Targowek, Warsaw
  - FutureMeds sp. z o. o., Wroclaw
- United Kingdom (7):
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrookes Hospital, Cambridge
  - Ninewells Hospital, Dundee
  - Northwick Park Hospital, Harrow
  - Hull Royal Infirmary - MAIN, Hull
  - Alder Hey Children's Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/